CLINICAL TRIAL: NCT04409379
Title: Association Between Relative Telomere Length and Severity of Cardiac Dysfunction
Brief Title: Association Between Telomere Length and Cardiac Dysfunction
Status: Completed | Type: Observational
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Lipeng Liu, Dr., Chinese Academy of Medical Sciences
Other Study IDs: YL2019100602
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Cardiac Toxicity; Acute Leukemia; Childhood Cancer
MeSH Terms: conditions — Cardiotoxicity; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Relative telomere length in peripheral blood cell
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- acute leukemia group: 300 patients were recruited, who have diagnosed with acute leukemia by bone marrow biopsy
  Interventions: Diagnostic Test: Relative telomere length

INTERVENTIONS:
Diagnostic Test: Relative telomere length — Relative telomere length in peripheral blood cell

SUMMARY:
Compelling epidemiological evidence indicates that alterations of relative telomere length (RTL) are associated with cardiac dysfunction caused by chemotherapy in children with acute leukemia (AL).The aim of this study was to explore association between RTL content in peripheral blood cells could be used as a risk predictor for severity of cardiac damage.

ELIGIBILITY:
Inclusion Criteria:

* 1. histological confirmed acute leukemia; 2. Preparing for chemotherapy;

Exclusion Criteria:

* 1.history of other malignancy; 2.blood transfusion within one month or prior bone marrow transplantation; 3.patients who reluctant to sign informed consent.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A total of 300 eligible acute leukemia patients were anticipated to include in this study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Relative telomere length | From date of admission until the date of discharging from hospital, assessed up to 5 days
  The ratio of RTL to hemoglobin contents was calculated for each sample from standard curves. After that, the ratio for each sample was normalized to a calibrator DNA in order to standardize between different runs, and then defined as the measurement of relative mtDNA contents.Relative expression of mtDNA were measured in young adults suffered from AL.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiao-Fan Zhu, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No